CLINICAL TRIAL: NCT01579903
Title: An Open-Label, Randomized, Two-period Crossover Study To Compare Relative Bioavailability of Two Formulations of Moroctocog Alfa (Af-cc) In Subjects With Moderately Severe Or Severe Hemophilia A (FVIII:C </=2%)
Brief Title: Relative Bioavailability Of Two Formulations Of Moroctocog Alfa (AF-CC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B1831077
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; moroctocog alfa (AF-CC); ReFacto AF; dual-chamber syringe; bioavailability
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects randomized to receive Treatment A during Period 1, then Treatment B during Period 2.
  Interventions: Drug: moroctocog alfa (AF-CC)
- Sequence 2 (Experimental): Subjects randomized to receive Treatment B during Period 1, then Treatment B during Period 2.
  Interventions: Drug: moroctocog alfa (AF-CC)

INTERVENTIONS:
Drug: moroctocog alfa (AF-CC) — Treatment A: 3000 IU moroctocog alfa (AF-CC) dual chamber syringe (including diluent); Treatment B: 1000 IU + 2000 IU moroctocog alfa (AF-CC) vials and separate diluent syringes
  Arms: Sequence 1
Drug: moroctocog alfa (AF-CC) — Treatment B: 1000 IU + 2000 IU moroctocog alfa (AF-CC) vials and separate diluent syringes; Treatment A: 3000 IU moroctocog alfa (AF-CC) dual chamber syringe (including diluent)
  Arms: Sequence 2

SUMMARY:
This study is being conducted to compare how moroctocog alfa (AF-CC) acts in the body when administered as 2 different dose presentations. The first is the current product vials with prefilled diluent syringes and the second is a new dual-chamber syringe dose presentation.

DETAILED DESCRIPTION:
This study is being conducted in order to satisfy a post-approval EMA commitment to compare the pharmacokinetics of the 2 dose presentations used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients at least 18 years old with severe or moderately severe hemophilia A (facto VIII concentration less than or equal to 2%).
* Negative test for facto VIII inhibitor.
* If applicable, HIV or hepatitis treatment is stable at the time of enrollment.
* Ability to abstain from use of FVIII products for 72 hours at a time.

Exclusion Criteria:

* History of any positive test result for factor VIII inhibitor.
* Presence of any bleeding disorder in addition to Hemophilia A.
* Body weight less than 50 kg.
* History of alcoholism.
* Treatment with investigational drug or device within 30 days prior to the Screening visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Single dose pharmacokinetics of moroctocog alfa (AF-CC) using noncompartmental analysis (primary PK parameters include: Cmax, AUClast, and AUCinf) | Periods 1 and 2, Day 1 through 4

SECONDARY OUTCOMES:
Single dose pharmacokinetics of moroctocog alfa (AF-CC) using noncompartmental analysis (secondary PK parameters include: tmax, λz, t1/2, CL, Vss, and FVIII Recovery) | Periods 1 and 2, Day 1 through Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Sofia, Bulgaria
- Pfizer Investigational Site, Budapest, Hungary
- Pfizer Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Shafer F, Charnigo RJ, Plotka A, Baumann J, Liang Y, Korth-Bradley J. Assessment of relative bioavailability of two presentations of moroctocog alfa (AF-CC) in subjects with moderately severe or severe hemophilia A. Clin Pharmacol Drug Dev. 2015 May-Jun;4(3):237-41. doi: 10.1002/cpdd.168. Epub 2014 Oct 27. PMID 27140804
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831077&StudyName=Relative%20Bioavailability%20Of%20Two%20Formulations%20Of%20Moroctocog%20Alfa%20%28AF-CC%29